CLINICAL TRIAL: NCT01269567
Title: Randomized Trial Comparing Drainage Versus no Drainage Following Rectal Excision With Low Anastomosis for Rectal Cancer
Brief Title: Drainage After Rectal Excision for Rectal Cancer
Acronym: GRECCAR 5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2010/24
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Rectal Cancer Surgery; Randomized Clinical Trial; Multicenter Study; Pelvic Drainage
Keywords: RectalNeoplasms; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases | interventions — Oviposition; Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drainage (Active Comparator): Rectal excision with aspiration pelvic drainage
  Interventions: Procedure: Laying and management of the drain (strictly randomized arm with drainage)
- No drainage (Experimental): Rectal excision without aspiration pelvic drainage
  Interventions: Procedure: No pelvic drainage

INTERVENTIONS:
Procedure: Laying and management of the drain (strictly randomized arm with drainage) — At the end of intervention, the surgeon will position an aspiration drain in order to permit a postoperative pelvic drainage. The drain will be positioned forward sacrum, behind anastomosis. The drain will be leaved in place between 3 and 5 days. The criteria of drain ablation are the absence of haemorrhagic liquid and/or un daily debit < 100ml. Nursing care will be daily with change of bottle for collect pelvic serosity, accounting of quantity of collected liquid and realization of a dried bandage through contact with penetration of the drain.
  Arms: Drainage
Procedure: No pelvic drainage — no aspiration drain at the end of intervention
  Arms: No drainage

SUMMARY:
After rectal excision, the rate of anastomotic leak and abscess is higher than after colic surgery. In order to limit and avoid the risk of pelvic sepsis after rectal excision, a prophylactic pelvic drainage is usually used. If current data have confirmed the uselessness of drainage in colic surgery, the question stay in abeyance in rectal surgery. This practice had never been evaluated in patients with rectal excision and low anastomosis (patients with a high risk of pelvic sepsis)

DETAILED DESCRIPTION:
After rectal excision, the rate of anastomotic leak and abscess is higher than after colic surgery. In order to limit and avoid the risk of pelvic sepsis after rectal excision, a prophylactic pelvic drainage is usually used. If current data have confirmed the uselessness of drainage in colic surgery, the question stay in abeyance in rectal surgery. This practice had never been evaluated in patients with rectal excision and low anastomosis (patients with a high risk of pelvic sepsis) The aim of the study is to assess the impact of pelvic drainage vs. non pelvic drainage on risk of pelvic sepsis after rectal excision for cancer with infraperitoneal anastomosis. The principal objective is to compare the rate of pelvic sepsis until 30 days between the 2 groups of patients who had a rectal excision with and without pelvic drainage. It is a randomized clinical trial of superiority, multicentric, without blinding, in 2 parallel groups with ratio (1:1): distribution of the number of patients in the groups.

ELIGIBILITY:
Inclusion Criteria:

* Rectal adenocarcinoma, histopathologically proved, with or without neoadjuvant treatment
* Stapler or manual infraperitoneal anastomosis
* With or without stoma
* With bowel preparation
* Open or laparoscopic approach
* Stage T1-T4 Nx Mx
* Age 18 years old or older
* Information of the patient and signature of informed consent
* Affiliation to a regime of social insurance

Exclusion Criteria:

* Colonic cancer (> 15 cm from anal verge)
* Abdominoperineal resection
* Associated resection (prostate, seminal bladder, vagina…)
* Simultaneous liver resection
* Total coloproctectomy
* Emergency
* Infected rectal tumour
* Pregnant women, suitable to be, or current suckling
* Persons deprived of freedom or under guardianship
* Persons under protection of justice
* Impossibility to accept the medical follow-up of the study for geographic , social or psychic reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pelvic sepsis | within the first 30 days after surgery
  Pelvic sepsis until 30 days after rectal excision is the primary end point. It is defined as the occurrence of an anastomotic leak revealed by peritonitis or discharge of gas, stools or pus, the vagina or the abdominal wound, and/or a pelvic abscess, between J0 and J30.

SECONDARY OUTCOMES:
Overall sepsis | up to 30 days after surgery
  Overall sepsis until 30 days (pelvic sepsis, wound abscess, urinary infection, pneumopathy, blood-poisoning)
Peri-operative mortality | up to 30 days after surgery
  Peri-operative mortality (hospital mortality and/or until 30 days after surgery if the patient is already going out of hospital)
Surgical morbidity according to Dindo classification | within the first 6 months after surgery
  Surgical morbidity according to Dindo classification
Re-surgery during the hospitalization | during the hospitalization
Rate of closure of stoma | within the first 6 months after surgery
  Rate of closure of stoma at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adélaïde Doussau, Dr, Study Chair — University Hospital, Bordeaux
Locations (22):
- France (22):
  - CHU d'AMIENS, Amiens
  - CH de BEAUVAIS, Beauvais
  - Service de Chirurgie Digestive - Hôpital Saint-André - CHU de Bordeaux, Bordeaux
  - Service de Chirurgie Générale et Digestive - Hôpital Beaujon, Clichy
  - Service de Chirurgie Digestive - Hôpital A. Michallon, La Tronche
  - APHP-Kremlin Bicetre, Le Kremlin-Bicêtre
  - Département de Chirurgie Oncologique - Centre Oscar Lambret, Lille
  - CHRU Lille, Lille
  - Centre Hospitalier Lyon Sud, Lyon
  - Département de Chirurgie Oncologique - Institut Paoli Calmette, Marseille
  - Service de Chirurgie Digestive et Viscérale - CHU Timone, Marseille
  - Département de Chirurgie Oncologique - CRLC Val d'Aurelle, Montpellier
  - Service de Chirurgie Digestive - CHU de Nantes - Hôtel Dieu, Nantes
  - Service de Chirurgie Générale et Digestive - Hôpital Saint-Antoine, Paris
  - APHP- Saint Joseph, Paris
  - Service de Chirurgie Digestive - Hôpital des Diaconnesses - La Croix Saint-Simon, Paris
  - CHU Poitiers, Poitiers
  - Service de Chirurgie Viscérale - CHU Pontchaillou, Rennes
  - Service de Chirurgie Digestive - CHU Charles Nicolle, Rouen
  - CHRU de Strasbourg, Strasbourg
  - Service de Chirurgie Digestive - Hôpital Purpan - Pavillon Dieulafoy, Toulouse
  - Service de Chirurgie Digestive et Générale - Brabois, Vandœuvre-lès-Nancy